CLINICAL TRIAL: NCT04918758
Title: Endoscopically-delivered Purastat for the Treatment of Haemorrhagic Radiation Proctopathy: a Randomised Feasibility Study
Brief Title: Endoscopically-delivered Purastat to Treat Bleeding Caused by Radiation Proctopathy
Acronym: PURASTAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B01152; 254308 (Other: IRAS)
Record Dates: First submitted 2021-05-13; First posted 2021-06-09 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Radiation Proctopathy
MeSH Terms: interventions — Water

STUDY DESIGN:
Intervention Model Description: Randomised to Purastat or treatment as usual (sucralfate enemas) using block sizes of 4 or 6, with block size itself determined at random. Randomisation will be stratified by Hospital
  Post-Market Phase
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Purastat Arm (Experimental): Purastat 5ml once monthly for 3 months
  Interventions: Device: Purastat Arm
- Standard Care Arm (Other): Sucralfate enemas 2g twice daily for 8 weeks
  Interventions: Drug: Standard Care Arm

INTERVENTIONS:
Device: Purastat Arm — Generic name of device and principal intended use(s):
  Still PuraStat from a CE mark perspective. PuraStat is an aqueous self-assembling peptide solution of 2.5% concentration RADA16
  Indication for use:
  PuraStat is indicated for haemostasis in the following situations encountered during surgery, when haemostasis by ligation or standard means is insufficient or impractical:
  * Bleeding from small blood vessels and oozing from capillaries of the parenchyma of solid organs. Oozing from vascular anastomoses
  * Bleeding from small blood vessels and oozing from capillaries of the GI tract following surgical procedures
  * Reduction of delayed bleeding following gastrointestinal endoscopic submucosal dissection (ESD) procedures in the colon.
  Other Names: PuraStat - 621-015
  Arms: Purastat Arm
Drug: Standard Care Arm — Sucralfate enemas 2g twice daily for 8 weeks, this is standard care in patients with haemorrhagic radiation proctopathy in the short term
  Other Names: Sucralfate enemas - Enemas of sucralfate suspension (2 gm in 20 ml water)
  Arms: Standard Care Arm

SUMMARY:
30,000 people in the UK are treated with pelvic radiotherapy each year. Rectal bleeding is a common symptom side effect caused by radiation proctopathy (RP). RP is due to the effect of radiation on the rectum (back passage) which causes poor blood supply (ischaemia) which leads to stiffness/scarring (fibrosis) and the development of abnormal blood vessels on the surface of the lining of the rectum (telangiectasia) which can bleed (1, 2). Six percent of patients will develop severe bleeding from RP (3), passing large amounts of blood and clots, often leading anaemia (low blood count) requiring either tablet or intravenous (IV) iron replacement, or blood transfusion.

There are very few safe, effective, evidence-based treatments available for RP. Purastat® is a new haemostatic agent (treatment that stops bleeding) which is licensed to treat bleeding from blood vessels in the gut. It is a liquid containing four peptides (protein building-blocks). When this liquid comes in contact with blood these peptides join together to form a mesh which closes the broken blood vessel thereby stopping the bleeding (4-7). Purastat is safe with no side effects and it breaks down amino acids, which are tissue building blocks that can be used to repair the site of injury (7). There are many studies which show that Purastat® is effective at stopping bleeding quickly and safely (within 10-20 seconds) (6-13). Early data from a case series of 21 patients by the research team has shown improvement in symptoms and endoscopic appearance. This study is a dual site randomised feasibility study of 80 patients. It will obtain initial data into the safety and efficacy Purastat in reducing bleeding in people with severe haemorrhagic RP. These data will be used to support funding for an definitive randomised controlled trial.

DETAILED DESCRIPTION:
Purastat is a new haemostatic agent (treatment that stops bleeding) which is licensed to treat bleeding from blood vessels in the gut. It is a liquid containing four peptides (protein building-blocks). When this liquid comes in contact with blood these peptides join together to form a mesh which closes the broken blood vessel thereby stopping the bleeding (4-7). Purastat is safe with no side effects and it breaks down amino acids, which are tissue building blocks that can be used to repair the site of injury (7). There are many studies which show that Purastat® is effective at stopping bleeding quickly and safely (within 10-20 seconds) (6-13). Early data from a case series of 21 patients by the research team has shown improvement in symptoms and endoscopic appearance.

Assessment Tools

1.Demographic data 2.7 day patient-reported rectal bleeding diary 3.Rectal bleeding score 4.Endoscopic grading: Zinicola score, rectal telangiectasia density score 5.Bloods: Haemoglobin concentration, ferritin 6.Blood transfusion requirement 7.Iron replacement requirement 8.Quality of life (EQ5D 5L) 9. Healthcare use including GP visits, hospital visit, A&E attendences, day case hospital visits, hospital admissions, blood transfusion and iron use.

The study duration will be 20 weeks (+/- 2 weeks). The timing of assessments will be baseline following consent (week 0); week 4 (+/- 1 week); week 8 (+/- 1 week); and week 20 (+/- 2 weeks).

Patients will be screened at their clinic appointment by study doctor. If they meet eligibility criteria, then verbal consent will be taken from the participant for the research nurse to contact them via telephone to discuss the study further. If the participant is happy to take part in the study following discussion with the research nurse then a follow-up telephone call will be arranged with study doctor for the participant to confirm happy to proceed and ask any further questions. An invitation letter plus participant information sheet and informed consent form will be either sent to the participant via post or email.

There are then 2 options for taking informed consent - either a telephone informed consent visit with return of informed consent to investigator site OR a face to face informed consent visit with respective study investigator and research nurse.

Demographic data plus details of cancer treatment, site, comorbidities, previous treatment for radiation proctopathy will be obtained. Participants will be allocated a study number and anonymised. They will then be randomised to Purastat or treatment as usual (sucralfate enemas) using block sizes of 4 or 6, with block size itself determined at random. Randomisation will be stratified by Hospital. An independent randomisation schedule will be generated for each of the Hospitals. Prescriptions for sucralfate 2g BD for 2 months will be issued to those randomised to treatment as usual for collection at first sigmoidoscopy appointment.

The research nurse will contact the participant to inform them of the arm they have been randomised to, confirm their baseline sigmoidoscopy visit date and ensure that they start completing their bleeding diary/healthcare utilisation starting 7 days before their baseline visit. Demographic data plus details of cancer treatment, site, comorbidities, previous treatment for radiation proctopathy will be obtained. Patients will be allocated a study number and anonymised. They will then be randomised to Purastat or treatment as usual (sucralfate enemas) using block sizes of 4 or 6, with block size itself determined at random.

Randomisation will be stratified by Hospital. An independent randomisation schedule will be generated for each of the Hospitals. Prescriptions for sucralfate 2g BD for 2 months will be issued to those randomised to treatment as usual for collection at first sigmoidoscopy appointment.

Week 0 -1 •The 7-day bleeding diary will be completed.

Week 0

* Patients will attend for first sigmoidoscopy.
* The bleeding diary will be collected and EORTC-QLQ-C30/EQ5D-5L/baseline healthcare utilisation questionnaire (covering the preceding 6 months including details of iron use and blood transfusion) completed.
* Baseline bloods will be taken (FBC, ferritin and iron studies).
* Assessment will be made using a rectal bleeding score.
* Sigmoidoscopy: insertion to rectum only to assess extent and severity of radiation proctopathy. Endoscopic images will be taken including in retroflexion. Endoscopic grading will be completed by the endoscopist. Images will be graded independently by a second gastroenterologist and any differences discussed and reviewed by a third if required.
* Purastat group: 5mls Purastat will be delivered.
* Treatment as usual group: sucralfate enemas collected from pharmacy: 2g BD for 8 weeks to start that day.
* The bleeding diary will be completed for the subsequent 7 days prior to their sigmoidoscopy visit.
* Next sigmoidoscopy visit is booked

Week 3

•The 7-day bleeding diary will be completed.

Week 4

* Patients will attend for second sigmoidoscopy.
* The bleeding diaries will be collected and EORTC-QLQ-C30/EQ5D-5L/baseline healthcare utilisation questionnaire (covering the preceding 4 weeks including details of iron use and blood transfusion) completed.
* Assessment will be made using a rectal bleeding score.
* Sigmoidoscopy: insertion to rectum only to assess extent and severity of radiation proctopathy. Endoscopic images will be taken including in retroflexion. Endoscopic grading will be completed by the endoscopist. Images will be graded independently by a second gastroenterologist and any differences discussed and reviewed by a third if required.
* 5mls Purastat will be delivered to those randomised into the Purastat group.
* The bleeding diary will be completed for the subsequent 7 days prior to their sigmoidoscopy visit.
* Next sigmoidoscopy visit is booked

Week 7 •The 7-day bleeding diary will be completed.

Week 8

* Patients will attend for third sigmoidoscopy.
* The bleeding diaries will be collected and EORTC-QLQ-C30/EQ5D-5L/baseline healthcare utilisation questionnaire (covering the preceding 4 weeks including details of iron use and blood transfusion) completed.
* Bloods will be taken (FBC, ferritin and iron studies).
* Assessment will be made using a rectal bleeding score.
* Sigmoidoscopy: insertion to rectum only to assess extent and severity of radiation proctopathy. Endoscopic images will be taken including in retroflexion. Endoscopic grading will be completed by the endoscopist. Images will be graded independently by a second gastroenterologist and any differences discussed and reviewed by a third if required.
* 5mls Purastat will be delivered to those randomised into the Purastat group.
* The bleeding diary will be completed for the subsequent 7 days prior to their sigmoidoscopy visit.
* Next sigmoidoscopy visit is booked

Week 19

•The 7-day bleeding diary will be completed.

Week 20

* Patients will attend for fourth sigmoidoscopy.
* The bleeding diaries will be collected and EORTC-QLQ-C30/EQ5D-5L/baseline healthcare utilisation questionnaire (covering the preceding 12 weeks including details of iron use and blood transfusion) completed.
* Bloods will be taken (FBC, ferritin and iron studies).
* Assessment will be made using a rectal bleeding score.
* Sigmoidoscopy: insertion to rectum only to assess extent and severity of radiation proctopathy. Endoscopic images will be taken including in retroflexion. Endoscopic grading will be completed by the endoscopist. Images will be graded independently by a second gastroenterologist and any differences discussed and reviewed by a third if required.
* CSQ-8 completed prior to discharge from the endoscopy unit
* End of patient involvement

Purastat delivery technique

* Insertion of sigmoidoscope into rectum
* Purastat will be spread over the telangiectasia using the designated catheter

On discharge from the endoscopy unit all patients will be given bleeding diaries and study team will arrange the next sigmoidoscopy appointment. Patients will be contacted by the research nurse via telephone at weeks 3, 7 and 19 to prompt completion of bleeding diary.

Individuals who dropped out of the study will be contacted by week 28 by the research nurse

ELIGIBILITY:
Inclusion criteria

* Age >16 years old
* Pelvic radiotherapy completed >6 months previously
* Endoscopically confirmed diagnosis of radiation proctopathy on lower GI endoscopy (sigmoidoscopy or colonoscopy) as characterised by the typical endoscopic appearances of superficial friable serpiginous telangiectasia, mucosal pallor and oedema
* Significant rectal bleeding (>weekly passage of blood into toilet bowl +/- anaemia which is ongoing for at least 3 months)
* Full colonic evaluation (colonoscopy or CT colonogram) to exclude other causes for rectal bleeding
* Capable of providing informed consent to a participant information sheet written in English

Exclusion criteria

* Age <16 years
* Unable to have full colonic evaluation to exclude other causes of rectal bleeding
* Other untreated cause for rectal bleeding
* Previous Purastat treatment for RP
* Previous Sucralfate treatment for RP

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility to deliver a full randomised controlled trial to determine if Purastat reduces lower gastrointestinal bleeding in patients with haemorrhagic radiation proctopathy in the short term compared to standard treatment with sucralfate enemas | through study completion, an average of 2 years
  Participants will be asked to describe their experience of the study process using a validated questionnaire (CSQ-8)
Feasibility to deliver a full randomised controlled trial to determine if Purastat reduces lower gastrointestinal bleeding in patients with haemorrhagic radiation proctopathy in the short term compared to standard treatment with sucralfate enemas | through study completion, an average of 2 years
  Participants will be asked to describe their reason for attrition verbally (end of study research nurse contact)
Feasibility to deliver a full randomised controlled trial to determine if Purastat reduces lower gastrointestinal bleeding in patients with haemorrhagic radiation proctopathy in the short term compared to standard treatment with sucralfate enemas | through study completion, an average of 2 years
  Attrition Rates to both study arms
Feasibility to deliver a full randomised controlled trial to determine if Purastat reduces lower gastrointestinal bleeding in patients with haemorrhagic radiation proctopathy in the short term compared to standard treatment with sucralfate enemas | through study completion, an average of 2 years
  rate of recruitment
Feasibility to deliver a full randomised controlled trial to determine if Purastat reduces lower gastrointestinal bleeding in patients with haemorrhagic radiation proctopathy in the short term compared to standard treatment with sucralfate enemas | through study completion, an average of 2 years
  Participants will be asked to describe their acceptability of the randomisation process verbally (end of study research nurse contact)
Feasibility to deliver a full randomised controlled trial to determine if Purastat reduces lower gastrointestinal bleeding in patients with haemorrhagic radiation proctopathy in the short term compared to standard treatment with sucralfate enemas | through study completion, an average of 2 years
  Participants will be asked to describe their acceptability of the recruitment process verbally (end of study research nurse contact)
Feasibility to deliver a full randomised controlled trial to determine if Purastat reduces lower gastrointestinal bleeding in patients with haemorrhagic radiation proctopathy in the short term compared to standard treatment with sucralfate enemas | through study completion, an average of 2 years
  Participants will be asked to describe their acceptability of the intervention on a validated questionnaire (CSQ-8)
Safety of endoscopically-delivered Purastat for the treatment of RP complicated by severe lower gastrointestinal bleeding. | through study completion, an average of 2 years
  Incidents of SAEs and AEs

SECONDARY OUTCOMES:
Usability of potential outcomes | through study completion, an average of 2 years
  Acceptability of questionnaires to participants (end of study research nurse contact)
Usability of potential outcomes | through study completion, an average of 2 years
  the best outcome measures will be the most clinically meaningful with the least missing data which show sufficient variation between patients, including determining whether there are floor/ceiling effects, and within patients over time on statistical analysis.
Usability of potential outcomes | through study completion, an average of 2 years
  The least data missing health economics outcome measures using validated questionnaires: EQ5D and health care utilisation questionnaire
To determine whether necessary information can be gathered | through study completion, an average of 2 years
  Percentage of missing data
To determine whether necessary information can be gathered | through study completion, an average of 2 years
  Attrition rates
Sample size determination for a definitive multicentre trial to determine the clinical and cost effectiveness of endoscopically-delivered Purastat for the treatment of RP complicated by severe lower gastrointestinal bleeding. | Completed 7 days before, 7 days after and Weeks 0, 4, 8 and 20 sigmoidoscopies
  Patient-reported bleeding episodes within the bleeding diary

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Henson, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Currently no- This may be updated in the future